CLINICAL TRIAL: NCT00102180
Title: Drug-Induced Sudden Death & Ventricular Arrhythmia
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sean Hennessy, Associate Professor of Epidemiology & of Pharmacology, University of Pennsylvania
Other Study IDs: 1287; 5R01HL076697 (NIH)
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases; Ventricular Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the relationship between the use of prescription drugs and the occurrence of ventricular arrhythmia and sudden death.

DETAILED DESCRIPTION:
BACKGROUND:

Drug-induced sudden cardiac death (also called sudden death, SD) and ventricular arrhythmia (VA) have arisen as major public health concerns in the last decade. Sudden death/ventricular arrhythmia have resulted in the withdrawal of more drugs in recent years than any other adverse drug reaction, and the identification of over 100 non-cardiac drugs as suspected of being high-risk. Unfortunately, controlled studies measuring the risks associated with specific drugs are very few in number, presumably because of the complexity of such studies and the massive sample sizes needed to study this outcome. Even studies in "large" databases have lacked adequate statistical power for crucial subgroup analyses. This lack of controlled data on clinical sudden death/ventricular arrhythmia has necessitated reliance on uncontrolled observations and on studies of putative markers of risk such as QTc prolongation in the electrocardiogram. However, the utility of uncontrolled observations is always subject to question, and the validity of these putative markers remains unknown. As a result, clinicians, patients, regulators, and drug manufacturers are ill-equipped to address the critical clinical and public health decisions concerning drug-induced sudden death/ventricular arrhythmia.

DESIGN NARRATIVE:

This study will compile a massive new pharmacoepidemiologic database of Medicaid data (linked with Medicare data for those enrolled in both programs, and with the Social Security Administration Death Masterfile) from five large Medicaid programs. This will be combined with the UK General Practice Research Database. This combined database will be used to conduct a series of nested case-control and case-crossover studies to measure the absolute and relative rate of all-cause death and sudden death/ventricular arrhythmia (SD/VA) associated with five of the most commonly used drug classes of greatest concern: antipsychotics, antidepressants, opioid analgesics, quinolone antibiotics, and macrolide antibiotics. A multi-stage investigative strategy will be used: Stage 1 will compile the database, assure its quality, and reproduce known associations. Stage 2a will compare drugs among the classes of interest. Stage 2b will use the case-crossover design to look for associations controlling for stable patient factors. Stage 2c will examine the effect of dose and inhibitors of pharmacokinetic clearance, the functional equivalent of high-dose use. Stage 3 will develop predictive indices to stratify patient subgroups receiving high-risk drugs.

ELIGIBILITY:
This combined database will be used to conduct a series of nested case-control and case-crossover studies to measure the absolute and relative rate of all-cause death and sudden death/ventricular arrhythmia (SD/VA) associated with five of the most commonly used drug classes of greatest concern: antipsychotics, antidepressants, opioid analgesics, quinolone antibiotics, and macrolide antibiotics.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medicaid enrollees from CA, FL, NY, OH and PA combined with the UK General Practice Research Database.
Sampling Method: Non-Probability Sample
Enrollment: 31000000 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
All cause death | All data years

SECONDARY OUTCOMES:
Composite outcome of sudden death and ventricular arrhythmia | All data years

CONTACTS AND LOCATIONS:
Overall Officials: Sean Hennessy, PharmD, PhD, Principal Investigator — University of Pennsylvania